CLINICAL TRIAL: NCT06107946
Title: The MuSt-PC: A Multidimensional Strategy to Improve Quality of Life of Patients With Multiple Symptoms and Palliative Care Needs - Pilot Study to Assess the Efficacy of a Clinical Decision Support System
Brief Title: The MuSt-PC: a Pilot Study to Assess Symptom Burden of Co-occuring Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11087
Record Dates: First submitted 2023-10-07; First posted 2023-10-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- symptom assessment (Other): Patients will have assessed symptom burden using the Dutch validated ESAS (called USD), build in the MuSt-PC tool. Thereafter, they will record symptom burden in a diary during 2 weeks.
  Interventions: Other: USD questionnaire

INTERVENTIONS:
Other: USD questionnaire — After a baseline screening symptom assessment, all eligible patients with at least 2 simultaneously occurring symptoms with a numeric rating score ≥4 on the 11 point scale on the Utrecht Symptom Diary, will be asked to fill out the Utrecht Symptom Diary during two weeks. In the first week twice daily (morning and evening), in the second week once daily (evening).

SUMMARY:
In this pilot study, physicians and nurse practitioners working in different care settings will use MuSt-PC, for adult patients with any life-limiting iilness, for whom the Surprise question is answered negatively: if the HCP answers "no" to the question "Would I be surprised if this patiënt died in the next 12 months?''. In total, at least 20 eligible patients will be recruited and asked to perform all study assessments.

DETAILED DESCRIPTION:
In this pilot study, physicians and nurse practitioners working in different care settings will use MuSt-PC, for adult patients with any life-limiting iilness, for whom the Surprise question is answered negatively: if the HCP answers "no" to the question "Would I be surprised if this patiënt died in the next 12 months?''. In total, at least 20 eligible patients will be recruited and asked to perform all study assessments.

After a baseline screening assessment, all eligible patients with at least 2 simultaneously occurring symptoms with a numeric rating score £4 on the 11 point scale on the Utrecht Symptom Diary, will be asked to fiil out the Utrecht Symptom Diary during two weeks.

In the first week twice daily (morning and evening), in the second week once daily (evening).

ELIGIBILITY:
Inclusion Criteria:

* Patients identified as in a palliative care trajectory (based on a negative answer to the surprise question "Would I be surprised if this patiënt died in the next 12 months?")
* All primary diseases (cancer, non-cancer (e.g. COPD, haart failure, frailty)
* Patients should have at least two symptoms on the Utrecht Symptom Diary with a numeric rating score of 4 or higher
* Life expectancy of at least 4 weeks
* Able to fill out Dutch questionnaires
* Informed consent

Exclusion Criteria:

* Patients who are unable or unwilling to self-assess their symptoms at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Ability and willingness of patients to complete follow-up assessments | after 2 weeks
  the percentage of patients who completed all questionnaires during follow-up

SECONDARY OUTCOMES:
Recruitment of patients; the number of patients that consented and those that declined participation, as well as number of eligible patients. | after 2 weeks
  % of patients
Adherence to advice by patients provided based on the MuSt-PC CDSS | after 2 weeks
  % of patients
Patient impressions of the MuSt-PC CDSS | after 2 weeks
  10 questions with a 4-point Likert scale
Time until symptom burden decreases after the use of the MuSt-PC CDSS based on the filled out Utrecht Symptom Diaries (days) | after 2 weeks
  in days
Feedback about the follow-up assessments within this pilot | after 2 weeks
  open questions

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - LUMC, Leiden